CLINICAL TRIAL: NCT06304909
Title: Effect of Intravenous Dexmedetomidine Versus Dexamethasone for Management of Repound Pain After Supraclavicular Brachial Plexus Block
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Sayed Mohamed Ahmed, Resident, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2080278
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries | interventions — Dexmedetomidine; Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine group will receive 0.5 mcg/kg (Experimental)
  Interventions: Drug: Dexmedetomidine injection
- Dexamethasone group will receive 8mg/kg (Experimental)
  Interventions: Drug: Dexmedetomidine injection
- Control group will receive equivalent volume of saline 0.9%. (Experimental)
  Interventions: Drug: Dexmedetomidine injection

INTERVENTIONS:
Drug: Dexmedetomidine injection — Dexmedetomidine group will receive 0.5 mcg/kg
  Other Names: Dexamethasone

SUMMARY:
Effect of intravenous dexmedetomidine versus dexamethasone for management of repound pain after supraclavicular brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20_60 years old

  * Patients with ASA clinical status I/II
  * Patients scheduled for peripheral nerve block for upper extremity surgery

Exclusion Criteria:

* 1) they refused to participate 2) had preexisting neuropathy of the surgical limb 3) hypersensitivity to amide anesthetic 4) significant pulmonary disease 5) coagulopathy 6) sepsis 7) infection at the block site 8) hypersensitivity to dexmedetomidine & dexamethasone

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The incidence of rebound pain. | 1year
  Rebound pain is defined as an increase from well-controlled to severe pain typically within 12_24 h of resolution of the nerve block.

CONTACTS AND LOCATIONS:
Overall Officials: Wesam Nashat Ali, Assistant professor, Study Director — Assistant professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolny M, Stasiowski MJ, Zuber M, Marciniak R, Chabierska E, Pluta A, Jalowiecki P, Byrczek T. Randomized, comparative study of the effectiveness of three different techniques of interscalene brachial plexus block using 0.5% ropivacaine for shoulder arthroscopy. Anaesthesiol Intensive Ther. 2017;49(1):47-52. doi: 10.5603/AIT.2017.0009. PMID 28362032
- [Background] Brattwall M, Jildenstal P, Warren Stomberg M, Jakobsson JG. Upper extremity nerve block: how can benefit, duration, and safety be improved? An update. F1000Res. 2016 May 18;5:F1000 Faculty Rev-907. doi: 10.12688/f1000research.7292.1. eCollection 2016. PMID 27239291
- [Background] Falgas N, Sanchez-Valle R, Bargallo N, Balasa M, Fernandez-Villullas G, Bosch B, Olives J, Tort-Merino A, Antonell A, Munoz-Garcia C, Leon M, Grau O, Castellvi M, Coll-Padros N, Rami L, Redolfi A, Llado A. Hippocampal atrophy has limited usefulness as a diagnostic biomarker on the early onset Alzheimer's disease patients: A comparison between visual and quantitative assessment. Neuroimage Clin. 2019;23:101927. doi: 10.1016/j.nicl.2019.101927. Epub 2019 Jul 5. PMID 31491836
- [Background] Hamilton DL. Rebound pain: distinct pain phenomenon or nonentity? Br J Anaesth. 2021 Apr;126(4):761-763. doi: 10.1016/j.bja.2020.12.034. Epub 2021 Feb 5. No abstract available. PMID 33551124
- [Background] Bhatia P, Metta R. Rebound pain: Undesired, yet unexplored. J Anaesthesiol Clin Pharmacol. 2022 Oct-Dec;38(4):527-528. doi: 10.4103/joacp.joacp_435_22. Epub 2022 Dec 26. No abstract available. PMID 36778810
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Result] Hong B, Oh C, Jo Y, Chung W, Park E, Park H, Yoon S. The Effect of Intravenous Dexamethasone and Dexmedetomidine on Analgesia Duration of Supraclavicular Brachial Plexus Block: A Randomized, Four-Arm, Triple-Blinded, Placebo-Controlled Trial. J Pers Med. 2021 Dec 1;11(12):1267. doi: 10.3390/jpm11121267. PMID 34945739